CLINICAL TRIAL: NCT06517186
Title: Myocardial Mechanisms in Heart Failure With Preserved Ejection Fraction (MM-HFpEF) A HeartShare Clinical Study
Brief Title: Myocardial Mechanisms in Heart Failure With Preserved Ejection Fraction
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Mayo Clinic (Other); Wake Forest University Health Sciences (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sanjiv Shah, Stone Endowed Professor of Medicine, Director of Research, Bluhm Cardiovascular Institute, Principal Investigator, HeartShare Data Translation Center, Northwestern University
Other Study IDs: 24-000688
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Cardiac tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFpEF: Participants with HFpEF
- Non-HFpEF: Participants without HFpEF

SUMMARY:
The purpose of this study is to identify changes in heart tissue structure and biological function in patients with heart failure by performing an endomyocardial biopsy (EMB or heart biopsy) during a right heart catheterization (RHC). The ultimate goal is to use this information to develop new treatments for heart failure.

ELIGIBILITY:
Inclusion Criteria:

* HFpEF criteria

  1. Age ≥30 years.
  2. Left ventricular ejection fraction ≥50% measured by echocardiography, CMR or MUGA (measured within one year + clinical stability)
  3. Definition of HFpEF: signs and/or symptoms of HF, NYHA functional class II-IV, and at least one of the following:

     1. Elevated BNP (≥75 pg/ml in sinus rhythm or ≥225 pg/ml in atrial fibrillation/flutter) or NTproBNP (≥225 pg/ml in sinus rhythm or ≥675 in atrial fibrillation/flutter) at baseline. Choice of BNP or NTproBNP is based on availability at each clinical center.
     2. Prior HF hospitalization (primary reason for the hospitalization is HF with elevated natriuretic peptide levels [using the thresholds listed above], requiring IV diuresis for HF, or pulmonary edema or pulmonary vascular congestion on chest radiography).
     3. Previously documented elevated pulmonary capillary wedge pressure (PCWP) at rest (≥15 mmHg) or during exercise (≥25 mmHg for supine exercise or PCWP/cardiac output ratio ≥2 mmHg/L/min for upright exercise).
     4. Elevated H2FPEF score69 (≥5) or HFA-PEFF70 score (≥5).

Suspected HFpEF criteria

1. Age ≥30 years.
2. Left ventricular ejection fraction ≥50% measured by echocardiography, CMR or MUGA (measured within one year + clinical stability)
3. Signs and/or symptoms of HF, NYHA functional class II-IV and all of the following:

   1. Does not meet BNP or NT-proBNP criteria for HFpEF (above)
   2. No prior HF hospitalization meeting HF criteria (above)
   3. No previous hemodynamic catheterization documentation of HF (as above)

Exclusion Criteria:

* 1. Inadequate echo or fluoroscopic images.

  2. Neck anatomy unfavorable for jugular venous cannulation

  3. Therapy with direct oral anticoagulants without cessation for a period (age, renal function, and agent specific) deemed adequate to normalize coagulation according to local clinical guidelines.

  4. Previous or ongoing therapy with warfarin with INR ≥ 1.6 measured day before or of EMB

  5. Platelet count < 50,000/ml

  6. Active bleeding or coagulation disorder

  7. Infection or fever

  8. Endocarditis

  9. Pregnancy

  10. Intracardiac thrombus

  11. RV Aneurysm

  12. Clinically significant tricuspid, pulmonary or aortic valve stenosis

  13. Tricuspid or pulmonary mechanical valve prosthesis

  14. Left bundle branch block

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over 30 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Heart Failure with Preserved Ejection Fraction (HFpEF) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Shah, MD, Principal Investigator — Northwestern University; Margaret Redfield, MD, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Mass General Brigham, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

DOCUMENTS (1):
  • Study Protocol (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT06517186/Prot_000.pdf